CLINICAL TRIAL: NCT06044727
Title: Comparative Evaluation Of the Restorative Capacity Of Marginal Gingiva Using MINST and Conventional Subgingival Instrumentation Involving RT1 Gingival Recession: A Randomized Controlled Clinical Trial
Brief Title: MINST Versus Conventional Subgingival Instrumentation In RT1 Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anjali Periodontics 2022
Record Dates: First submitted 2023-09-08; First posted 2023-09-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): After phase 1 therapy, management of RT1 cases will be done with Minimally invasive non surgical periodontal therapy.
  Interventions: Procedure: Minimally invasive non surgical periodontal therapy
- Control Group (Active Comparator): After phase 1 therapy, management of RT1 cases will be done with Conventional subgingival instrumentation.
  Interventions: Procedure: Conventional subgingival instrumentation

INTERVENTIONS:
Procedure: Minimally invasive non surgical periodontal therapy — using Magnifying loupes
  Arms: Test group
Procedure: Conventional subgingival instrumentation — Conventional subgingival instrumentation
  Arms: Control Group

SUMMARY:
Gingival recession is a common condition and its extent and prevalence increase with age. Majority of patients probably present with localized and shallow gingival recession that need a specific treatment because they are susceptible to further apical displacement of gingival margin. So if gingival recession is detected early, removal of causative factors and non surgical treatments initiated then it can prevent more advanced mucogingival defects. Studies have shown that non surgical periodontal therapy including proper oral hygiene instructions, periodic scaling and root planning obtained successful root coverage in shallow gingival recession. Minimal invasive non surgical periodontal therapy (MINST)uses the delicate instruments and magnifying loupes performing periodontal debridement with more effective calculus and biofilm removal and less soft tissue trauma , maintain the tissue architecture, benefit the healing phase, improve the clinical results and increase visibility. There is no study to evaluate efficacy of MINST versus conventional subgingival instrumentation in the restorative capacity of marginal gingival in RT1 gingival recession , so the present study will be conducted to compare and evaluate the efficacy of minimal invasive non surgical periodontal therapy (MINST) and conventional subgingival instrumentation in the restorative capacity of marginal gingiva involving RT1 gingival recession.

DETAILED DESCRIPTION:
TITLE:

"Comparative Evaluation Of the Restorative Capacity Of Marginal Gingiva Using Minimal Invasive Non-Surgical Periodontal Therapy and Conventional Subgingival Instrumentation Involving RT1 Gingival Recession : A Randomized controlled clinical trial."

RATIONALE:

Gingival recession is a common condition and its extent and prevalence increase with age. Majority of patients probably present with localized and shallow gingival recession that need a specific treatment because they are susceptible to further apical displacement of gingival margin. So if gingival recession is detected early, removal of causative factors and non surgical treatment initiated then it can prevent more advanced mucogingival defects. Studies have shown that non surgical periodontal therapy including proper oral hygiene instructions, periodic scaling and root planning obtained successful root coverage in shallow gingival recession. Minimal invasive non surgical periodontal therapy (MINST)uses the delicate instruments and magnifying loupes performing periodontal debridement with more effective calculus and biofilm removal and less soft tissue trauma , maintain the tissue architecture, benefit the healing phase, improve the clinical results and increase visibility. There is no study to evaluate efficacy of MINST versus conventional subgingival instrumentation in the restorative capacity of marginal gingival in RT1 gingival recession , so the present study will evaluate the same.

AIM:

To compare and evaluate the efficacy of minimal invasive non surgical periodontal therapy (MINST) and conventional subgingival instrumentation in the restorative capacity of marginal gingiva involving RT1 gingival recession.

OBJECTIVES:

PRIMARY OBJECTIVE

1. Comparative evaluation of improvement in recession depth, recession width and root coverage percentage after using Conventional Subgingival Instrumentation.
2. Comparative evaluation of improvement in recession depth, recession width and root coverage percentage after using MINST.

SECONDARY OBJECTIVE To assess the improvement in other clinical parameters which include- Clinical attachment level (CAL), Probing Pocket Depth (PPD), Bleeding on probing (BOP), Plaque index (PI), Gingival index (GI),Gingival thickness (GT), Keratinized tissue width (KTW) and Visual analog scale for patient reported outcome of pain and hypersensitivity.

SETTING:

Department of Periodontics and Oral Implantology, PGIDS, Rohtak, Haryana.

STUDY DESIGN:

Randomized controlled clinical trial

TIME FRAME:

12-14 months

POPULATION:

Systemically healthy patients with RT1 gingival recession will be recruited in the study from out patient department of Periodontology. Recruitment of the patients for the study will be based on eligibility criteria after obtaining informed and written consent.

MATERIAL AND METHOD:

Systemically healthy patients having RT1 gingival recession will be assigned into control group (Conventional subgingival instrumentation) and test group( MINST). One group will be treated with Conventional subgingival instrumentation and other group will be treated with MINST. All the patients will be recalled twice in 1st and 2nd month followed by 3 months and 6 months for reevaluation. Standardized oral hygiene instructions will be imparted and reinforced at each appointment. Minimal Invasive non surgical periodontal therapy(MINST) and conventional subgingival instrumentation will be performed at follow up visits if required.

STATISTICAL ANALYSIS:

Data recorded will be processed by standard statistical analysis. The normality of distribution of data will be examined by Shapiro Wilk test. Statistical analysis will be performed according to distribution of data. If it is in normal distribution, inter group comparison will be done by using Independent T test and paired T test will be use for intragroup comparison and if non normal distribution of data, inter group comparison will be done by Mann-whitney U test and intragroup by signed rank test . The Chi square test will be applied to analyze categoric data. Correlation and association between predictors and dependent variables will be analyzed by correlation analysis and regression analysis.

RESEARCH QUESTION:

Does the use of minimal invasive non surgical periodontal therapy enhances the restorative capacity of marginal gingiva of RT1 gingival recession than conventional subgingival instrumentation.

P- POPULATION: systemically healthy patients with RT1 gingival recession

I- INTERVENTION: Conventional subgingival instrumentation with RT1 gingival recession

C-COMPARATOR: Minimal invasive non surgical periodontal therapy with RT1 gingival recession O- OUTCOME: Changes in recession depth, recession width and root coverage percentage.

T- TIME: 12-14 months

F- Feasibility: adequate sample size, infrastructure, time , study design.

I- Interesting: as it will be using minimal invasive non surgical periodontal therapy in RT1 gingival recession.

N- Novelty: no study was found in literature comparing the effects of minimal invasive non surgical periodontal therapy and conventional subgingival instrumentation in RT1 shallow gingival recession.

E- Ethical: Ethical

R- Relevant: exploring the efficacy of minimal invasive non surgical periodontal therapy and conventional subgingival instrumentation in RT1 gingival recession.

ELIGIBILITY:
Inclusion Criteria:

1. Gingival Recession Type 1(RT1) by Cairo et al 2011in esthetic zone including maxillary and mandibular anteriors and premolars, otherwise systemically healthy
2. Gingival Recession ≤3mm associated with plaque induced inflammation and identifiable CEJ
3. Age 20 years to 50 years
4. Providing a written and verbal informed consent.

Exclusion Criteria:

1. Patient with systemic disease that can influence the outcome of therapy.
2. Pregnant females or on oral contraceptive pills or hormone replacement therapy.
3. Smokers and patients undergoing orthodontic therapy
4. Physically and mentally impaired patients.
5. Non vital, mal-positioned tooth
6. Presence of cervical abrasions or restorations in the area
7. Previous history of periodontal surgery on the involved sites.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Recession Depth | 6 months
  recorded in mm with a periodontal probe from the cementoenamel junction to the crest of the gingival margin at mid labial region.
Recession Width | 6 months
  recorded in mm with a periodontal probe from the mesial to distal gingival margin at the level of cementoenamel junction.
Root Coverage % | 6 months
  Will be calculated according to the formula Root Coverage percentage =Recession depth(preop -postop)*100/Recession depth preoperative

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Yadav, BDS, Principal Investigator — Postgraduate Institute of Dental Sciences Rohtak
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No